CLINICAL TRIAL: NCT07381088
Title: The Effect of Education Provided in Primary Health Care Services on Vaccine Hesitancy, Digital Vaccine Literacy, Eco-Anxiety, and Perceived Vulnerability to Diseases Among Parents of Children Aged 0-2 Years
Brief Title: Effect of Primary Care Education on Parents' Health-Related Perceptions and Attitudes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Muhammet Faruk Yigit, Assistant Professor / Dr., Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12.01.2026-228398
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Vaccine Hesitancy; Health Education; Digital Health Literacy; Eco-anxiety; Vulnerability to Disease; Childhood Immunization
Keywords: Primary Health Care; Family Health Center; Parents; Children aged 0-2 years; Structured education program; Pretest-posttest; Misinformation; Health beliefs
MeSH Terms: conditions — Vaccination Hesitancy; Health Education; Communication

STUDY DESIGN:
Intervention Model Description: This study uses a quasi-experimental, pre-test-post-test, parallel-group design with an intervention group and a control group. Participants are assigned to either a structured education program delivered in primary health care settings or to routine care without additional education.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Structured Education (Experimental): Participants assigned to this arm will receive a structured, face-to-face education program delivered in a primary health care setting. The program consists of three weekly sessions, each lasting approximately 30-40 minutes. The education covers childhood vaccination, vaccine hesitancy, digital vaccine literacy, eco-anxiety, and perceived vulnerability to diseases.
  Interventions: Behavioral: Structured Education Program
- Arm Type: Control Group (No Intervention) (No Intervention): Participants assigned to this arm will receive routine services provided by the Family Health Center. No additional educational intervention will be administered during the study period.

INTERVENTIONS:
Behavioral: Structured Education Program — A structured education program consisting of three face-to-face sessions delivered once per week in a primary health care setting. Each session lasts approximately 30-40 minutes and focuses on childhood vaccination, vaccine hesitancy, digital vaccine literacy, eco-anxiety, and perceived vulnerability to diseases.
  Arms: Arm 1 (Experimental): Structured Education

SUMMARY:
This study aims to evaluate the effect of a structured education program delivered in primary health care settings on parents of children aged 0-2 years. The education focuses on childhood vaccination and related health perceptions.

Parents will receive education covering childhood vaccines, vaccine hesitancy, evaluation of vaccine-related information obtained from digital sources, eco-anxiety, and perceived vulnerability to diseases. The study examines whether this education influences parents' levels of vaccine hesitancy, digital vaccine literacy, eco-anxiety, and perceived vulnerability to diseases. The findings are expected to contribute to the development of effective educational interventions in primary health care services to support informed parental decision-making regarding childhood vaccination.

DETAILED DESCRIPTION:
Childhood vaccination is one of the most effective and cost-efficient public health interventions for preventing infectious diseases. However, vaccine hesitancy among parents has emerged as a significant public health concern, particularly in the context of misinformation disseminated through digital media. Parents' attitudes toward vaccination are influenced not only by face-to-face communication with health professionals but also by their ability to access, evaluate, and use vaccine-related information from online sources. In addition, environmental concerns and climate-related health risks have increased levels of eco-anxiety, which may influence individuals' perceptions of vulnerability to diseases and health-related decision-making.

This study is designed as a quasi-experimental, pre-test-post-test, control-group study to evaluate the effect of a structured education program delivered in primary health care services on parents of children aged 0-2 years. The study will be conducted at a Family Health Center in Van, Türkiye. Parents who meet the inclusion criteria and provide written informed consent will be enrolled in the study.

Participants will be assigned to either an intervention group or a control group. Parents in the intervention group will receive a structured education program consisting of three face-to-face sessions delivered once per week, with each session lasting approximately 30-40 minutes. The education program includes: (1) childhood vaccines, vaccine hesitancy, and common misconceptions; (2) digital vaccine literacy, reliable information sources, and coping with misinformation; and (3) eco-anxiety, environmental health concerns, perceived vulnerability to diseases, and coping strategies. The control group will receive routine services provided by the Family Health Center and will not receive any additional educational intervention.

Data will be collected using validated self-report instruments administered before the intervention and 15 days after completion of the final education session. The primary outcomes include changes in vaccine hesitancy, digital vaccine literacy, eco-anxiety, and perceived vulnerability to diseases. Sociodemographic information will also be collected. All data will be collected through face-to-face interviews in a private setting, and participant confidentiality will be ensured by using coded identifiers instead of personal information.

The study aims to determine whether education provided within primary health care services can effectively improve parents' attitudes and perceptions related to vaccination and child health. The results are expected to inform future public health education strategies targeting parents during early childhood.

ELIGIBILITY:
Inclusion Criteria:

* Parents who have at least one child aged 0-2 years
* Attendance at the Van Tuşba Family Health Center
* Ability to read and write in Turkish
* Willingness to participate voluntarily in the study
* Provision of written informed consent

Exclusion Criteria:

* Individuals with a diagnosed psychiatric disorder
* Individuals with cognitive or sensory impairments that prevent effective communication
* Individuals who are unable to attend the education sessions
* Individuals who do not complete the baseline assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Vaccine Hesitancy Level | Baseline (pre-intervention) and 15 days after completion of the education program
  Change in parents' level of vaccine hesitancy measured using the Parent Vaccine Hesitancy Scale.
  The scale consists of 10 items and 2 subdimensions, with items 1, 2, 3, 4, 6, and 7 reverse-coded. It includes the Lack of Confidence subdimension (items 1, 2, 3, 4, 6, 7, and 8) and the Risks subdimension (items 5, 9, and 10). The scale is rated on a five-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree), and the total score is calculated by summing the item scores; higher total scores indicate lower levels of vaccine hesitancy.
Digital Vaccine Literacy Level | Baseline and 15 days after completion of the education program
  Change in parents' digital vaccine literacy level measured using the Digital Vaccine Literacy Scale.
  The scale consists of a total of 7 items and 3 subdimensions: trust in and understanding of official information (items 1-2), trust in and understanding of information on social media (items 3-4), and evaluation and application of online vaccine information (items 5-7). Each item is rated on a four-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree). The total score ranges from 7 to 28, with higher scores indicating a higher level of digital vaccine literacy.
Eco-Anxiety Level | Baseline and 15 days after completion of the education program
  Change in parents' eco-anxiety level measured using the Hogg Eco-Anxiety Scale (HEAS-13) The scale consists of 13 items and four subdimensions (anxiety symptoms, rumination, behavioral symptoms, and concern about personal impact), with each item rated on a five-point Likert scale (0 = not at all, 1 = some days, 2 = most days, 3 = nearly every day). Higher scores on the scale indicate higher levels of eco-anxiety.
Perceived Vulnerability to Disease | Baseline and 15 days after completion of the education program
  Change in parents' perceived vulnerability to disease measured using the Perceived Vulnerability to Disease Scale.
  The scale consists of a total of 15 items and two subdimensions: Perceived Infectability (items 2, 5, 6, 8, 10, 12, and 14) and Germ Aversion (items 1, 3, 4, 7, 9, 11, 13, and 15). Items 3, 5, 11, 12, 13, and 14 are reverse-scored. The total score obtainable from the scale ranges from 7 to 105. The scale is structured as a seven-point Likert type, ranging from 1 (strongly disagree) to 7 (strongly agree), and higher scores indicate a higher perceived vulnerability to diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yuzuncu Yil University, Van, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical considerations and the absence of explicit consent for data sharing in the informed consent process. Data will be used only for the purposes of the present study and reported in aggregate form to ensure participant confidentiality.

REFERENCES:
- [Result] Betsch C, Brewer NT, Brocard P, et al. Opportunities and challenges of Web 2.0 for vaccination decisions. Vaccine. 2018;36(25):3727-3733. doi:10.1016/j.vaccine.2018.02.025
- [Result] World Health Organization. Ten threats to global health in 2019. World Health Organization; 2019. https://www.who.int/news-room/spotlight/ten-threats-to-global-health-in-2019